CLINICAL TRIAL: NCT06956885
Title: Maintenance or Withdrawal of Urate Lowering Therapy According to Ultrasound Features in Gout Patients: a Randomised Controlled Trial
Brief Title: Maintenance or Withdrawal of Urate Lowering Therapy According to Ultrasound Features in Gout Patients: a Randomised Controlled Trial Stop Treatment In Gout
Acronym: STING
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: APHP230854
Record Dates: First submitted 2025-04-25; First posted 2025-05-04 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-04

CONDITIONS: Gout Chronic

STUDY DESIGN:
Intervention Model Description: Multicentre, parallel arm, non-blinded randomised controlled non-inferiority clinical trial. Gout patients in remission and no urate deposits as assessed by US will be randomised to i) a maintenance group -ULT will be pursued - or ii) a withdrawal experimental group - discontinuation of ULT -.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Discontinuation of urate lowering therapy (Experimental)
  Interventions: Drug: Discontibuation of oral ULT
- Continuation of urate lowering therapy (usual care) (Active Comparator)
  Interventions: Drug: Maintenance of ULT

INTERVENTIONS:
Drug: Discontibuation of oral ULT — Patients will stop the ULT at D0. They will have an US scan to look for urate deposits at each visit.
  Arms: Discontinuation of urate lowering therapy
Drug: Maintenance of ULT — Patients will continue their ULT according to the recommendations of the Eular and French Society of Rheumatology, to maintain their SUA levels below 60 mg/l.
  Arms: Continuation of urate lowering therapy (usual care)

SUMMARY:
According to international recommendations, urate lowering therapy (ULT), mainly the xanthine oxidase inhibitors (XOIs) allopurinol and febuxostat, should be prescribed lifelong in gout patients. However, this recommendation comes up against very poor adherence to ULT, since around half of patients stop their treatment at 5 years. Moreover, there is uncertainty about the cardiovascular tolerance of febuxostat taken over the long term. Finally, although XOIs are generally well tolerated, they can cause side effects and require regular biological monitoring. The hypothesis is that the risk of flares following withdrawal of ULT is very low in gout patients when urate store is depleted and repeated ultrasounds (US) do not demonstrate the reappearance of urate deposits.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Gout, defined according to the 2015 ACR/EULAR classification criteria
* No flares for at least 2 years
* No tophi
* Currently receiving allopurinol or febuxostat taken for at least 2 years and SUA levels ≤ 60 mg/l
* No urate deposit on ultrasound at inclusion visit at both MTPs 1 and knees
* Ability to provide informed consent
* Women of childbearing potential (WOCBP) are required to have a negative pregnancy test before treatment and must agree to maintain during treatment highly effective contraception (ie,abstinence, combined estrogen- and progestogen-containing hormonal contraception, ovulation inhibitors (Oral, Intravaginal, Transdermal); Progestogen-only hormonal contraception associated with inhibition of ovulation (Oral, Injectable, Implantable); Intrauterine device (IUD); Intrauterine hormone-releasing system (IUS); Bilateral tubal occlusion; Vasectomised partner).
* Health Insurance

Exclusion Criteria:

* Unstable systemic medical condition (e.g., New York Heart Association stage IV heart failure, recent myocardial infarction, advanced cancer)
* History of allergy to allopurinol or febuxostat or one of the excipients
* Association with azathioprine, mercaptopurine (cytostatics-antimetabolites)
* Contraindications to experimental medicinal products or auxiliary medicinal products
* CKD stage 4 (eGFR less than 30 ml/mn/1.73 m2)
* Ongoing treatment with uricosurics (benzbromarone and probenecid) or uricase
* Patient on SMA (state medical aid-AME)
* Participation in other clinical trial on medicinal product for human use
* Lack of contraception for women of childbearing potential.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2029-05-01 (Estimated); Study Completion 2030-05-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients experiencing one or more flares | At 2 years
  According to the Gaffo's criteria

SECONDARY OUTCOMES:
Proportion of patients experiencing one or more flares | At 6 months
  According to both the Gaffo's criteria and the patient-reported Gout Attack Intensity Score (GAIS)
Proportion of patients experiencing one or more flares | At 12 months
  According to both the Gaffo's criteria and the patient-reported Gout Attack Intensity Score (GAIS)
Proportion of patients experiencing one or more flares | At 18 months
  According to both the Gaffo's criteria and the patient-reported Gout Attack Intensity Score (GAIS)
Proportion of patients experiencing one or more flares | At 30 months
  According to both the Gaffo's criteria and the patient-reported Gout Attack Intensity Score (GAIS)
Proportion of patients experiencing one or more flares | At 36 months
  According to both the Gaffo's criteria and the patient-reported Gout Attack Intensity Score (GAIS)
Mean flare rates | At 6 months
  According to both the Gaffo's criteria and the patient-reported Gout Attack Intensity Score (GAIS)
Mean flare rates | At 12 months
  According to both the Gaffo's criteria and the patient-reported Gout Attack Intensity Score (GAIS)
Mean flare rates | At 18 months
  According to both the Gaffo's criteria and the patient-reported Gout Attack Intensity Score (GAIS)
Mean flare rates | At 24 months
  According to both the Gaffo's criteria and the patient-reported Gout Attack Intensity Score (GAIS)
Mean flare rates | At 30 months
  According to both the Gaffo's criteria and the patient-reported Gout Attack Intensity Score (GAIS)
Mean flare rates | At 36 months
  According to both the Gaffo's criteria and the patient-reported Gout Attack Intensity Score (GAIS)
US features of gout at MPT1s | At 6 months
  Double contour sign, tophi, aggregates for withdrawal arm
US features of gout at MPT1s | At 12 months
  Double contour sign, tophi, aggregates for withdrawal arm
US features of gout at MPT1s | At 18 months
  Double contour sign, tophi, aggregates for withdrawal arm
US features of gout at MPT1s | At 24 months
  Double contour sign, tophi, aggregates for both arms
US features of gout at MPT1s | At 30 months
  Double contour sign, tophi, aggregates for withdrawal arm
US features of gout at MPT1s | At 36 months
  Double contour sign, tophi, aggregates for withdrawal arm
US features of gout at knees | At 6 months
  Double contour sign for withdrawal arm
US features of gout at knees | At 12 months
  Double contour sign for withdrawal arm
US features of gout at knees | At 18 months
  Double contour sign for withdrawal arm
US features of gout at knees | At 24 months
  Double contour sign for both arms
US features of gout at knees | At 30 months
  Double contour sign for withdrawal arm
US features of gout at knees | At 36 months
  Double contour sign for withdrawal arm
Urate levels | At 6 months
Urate levels | At 12 months
Urate levels | At 18 months
Urate levels | At 24 months
Urate levels | At 30 months
Urate levels | At 36 months
Change from baseline of patient's global assessment of disease activity | At 12 months
  Outcome Measures in Rheumatology (OMERACT) core outcome domains for long-term gout studies 0-5-point Likert scale, the higher the score the more severe the disease
Change from baseline of patient's global assessment of disease activity | At 24 months
  Outcome Measures in Rheumatology (OMERACT) core outcome domains for long-term gout studies 0-5-point Likert scale, the higher the score the more severe the disease
Change from baseline of patient's global assessment of disease activity | At 36 months
  Outcome Measures in Rheumatology (OMERACT) core outcome domains for long-term gout studies 0-5-point Likert scale, the higher the score the more severe the disease
Change from baseline in Healthrelated quality of life | At 12 months
  Outcome Measures in Rheumatology (OMERACT) core outcome domains for long-term gout studies EuroQol 5-domain-3L (EQ-5D3L) questionnaire The QLQ-C30 is composed of both multi-item scales and single-item measures. These include five functional scales, three symptom scales, a global health status / QoL scale, and six single items. Each of the multi-item scales includes a different set of items - no item occurs in more than one scale. All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level. A high score for a functional scale represents a high/healthy level of functioning. A high score for the global health status/ QoL represents a high QoL and a high score for a symptom scale/item represents a high level of symptomatology/problems
Change from baseline in Healthrelated quality of life | At 24 months
  Outcome Measures in Rheumatology (OMERACT) core outcome domains for long-term gout studies EuroQol 5-domain-3L (EQ-5D3L) questionnaire The QLQ-C30 is composed of both multi-item scales and single-item measures. These include five functional scales, three symptom scales, a global health status / QoL scale, and six single items. Each of the multi-item scales includes a different set of items - no item occurs in more than one scale. All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level. A high score for a functional scale represents a high/healthy level of functioning. A high score for the global health status/ QoL represents a high QoL and a high score for a symptom scale/item represents a high level of symptomatology/problems
Change from baseline in Healthrelated quality of life | At 36 months
  Outcome Measures in Rheumatology (OMERACT) core outcome domains for long-term gout studies EuroQol 5-domain-3L (EQ-5D3L) questionnaire The QLQ-C30 is composed of both multi-item scales and single-item measures. These include five functional scales, three symptom scales, a global health status / QoL scale, and six single items. Each of the multi-item scales includes a different set of items - no item occurs in more than one scale. All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level. A high score for a functional scale represents a high/healthy level of functioning. A high score for the global health status/ QoL represents a high QoL and a high score for a symptom scale/item represents a high level of symptomatology/problems
Change from baseline in Activity limitation | At 12 months
  Outcome Measures in Rheumatology (OMERACT) core outcome domains for long-term gout studies Health Assessment Questionnaire II is a 10-item score. Each item is rated on a 4-point Likert scale HAQ-II mean score ranges from 0 (no disability) to 3 (severe disability)
Change from baseline in Activity limitation | At 24 months
  Outcome Measures in Rheumatology (OMERACT) core outcome domains for long-term gout studies Health Assessment Questionnaire II is a 10-item score. Each item is rated on a 4-point Likert scale HAQ-II mean score ranges from 0 (no disability) to 3 (severe disability)
Change from baseline in Activity limitation | At 36 months
  Outcome Measures in Rheumatology (OMERACT) core outcome domains for long-term gout studies Health Assessment Questionnaire II is a 10-item score. Each item is rated on a 4-point Likert scale HAQ-II mean score ranges from 0 (no disability) to 3 (severe disability)
Incidence of Major CardioVascular events | At 6 months
  Including nonfatal stroke, nonfatal myocardial infarction, cardiovascular death
Incidence of Major CardioVascular events | At 12 months
  Including nonfatal stroke, nonfatal myocardial infarction, cardiovascular death
Incidence of Major CardioVascular events | At 18 months
  Including nonfatal stroke, nonfatal myocardial infarction, cardiovascular death
Incidence of Major CardioVascular events | At 24 months
  Including nonfatal stroke, nonfatal myocardial infarction, cardiovascular death
Incidence of Major CardioVascular events | At 30 months
  Including nonfatal stroke, nonfatal myocardial infarction, cardiovascular death
Incidence of Major CardioVascular events | At 36 months
  Including nonfatal stroke, nonfatal myocardial infarction, cardiovascular death
estimated glomerular filtration rate (eGFR) | At 6 months
  Renal function
estimated glomerular filtration rate (eGFR) | At 12 months
  Renal function
estimated glomerular filtration rate (eGFR) | At 18 months
  Renal function
estimated glomerular filtration rate (eGFR) | At 24 months
  Renal function
estimated glomerular filtration rate (eGFR) | At 30 months
  Renal function
estimated glomerular filtration rate (eGFR) | At 36 months
  Renal function
Incidence of comorbidities | At 12 months
  Charlson index Total score varies from 0 to >=5 The lower the score the higher the estimated 10-year survival
Incidence of comorbidities | At 24 months
  Charlson index Total score varies from 0 to >=5 The lower the score the higher the estimated 10-year survival
Incidence of comorbidities | At 36 months
  Charlson index Total score varies from 0 to >=5 The lower the score the higher the estimated 10-year survival
Overall Survival | At 12 months
Overall Survival | At 24 months
Overall Survival | At 36 months
Consumption of other drugs | At 6 months
  Colchicine, NSAIDs, steroids using a patient self-reported notebook
Consumption of other drugs | At 12 months
  Colchicine, NSAIDs, steroids using a patient self-reported notebook
Consumption of other drugs | At 18 months
  Colchicine, NSAIDs, steroids using a patient self-reported notebook
Consumption of other drugs | At 24 months
  Colchicine, NSAIDs, steroids using a patient self-reported notebook
Consumption of other drugs | At 30 months
  Colchicine, NSAIDs, steroids using a patient self-reported notebook
Consumption of other drugs | At 36 months
  Colchicine, NSAIDs, steroids using a patient self-reported notebook
Incidence of adverse events and serious adverse events | At 6 months
  According to CTCAE v5.0 classification (Common Terminology Criteria for Adverse Events)
Incidence of adverse events and serious adverse events | At 12 months
  According to CTCAE v5.0 classification (Common Terminology Criteria for Adverse Events)
Incidence of adverse events and serious adverse events | At 18 months
  According to CTCAE v5.0 classification (Common Terminology Criteria for Adverse Events)
Incidence of adverse events and serious adverse events | At 24 months
  According to CTCAE v5.0 classification (Common Terminology Criteria for Adverse Events)
Incidence of adverse events and serious adverse events | At 30 months
  According to CTCAE v5.0 classification (Common Terminology Criteria for Adverse Events)
Incidence of adverse events and serious adverse events | At 36 months
  According to CTCAE v5.0 classification (Common Terminology Criteria for Adverse Events)
Adherence to ULT | At 6 months
  Assessed by a questionnaire
Adherence to ULT | At 12 months
  Assessed by a questionnaire
Adherence to ULT | At 18 months
  Assessed by a questionnaire
Adherence to ULT | At 24 months
  Assessed by a questionnaire
Adherence to ULT | At 30 months
  Assessed by a questionnaire
Adherence to ULT | At 36 months
  Assessed by a questionnaire
Incremental Cost effectiveness ratios estimating cost per QALY gained | Up to 36 months
Incremental Cost effectiveness ratios estimating cost per flare avoided. | Up to 36 months

IPD SHARING:
Plan to Share IPD: Undecided